CLINICAL TRIAL: NCT01795274
Title: Phase I Study Evaluating the Treatment of Patients With Locally Advanced Pancreatic Cancer With Carbon Ion Radiotherapy: The PHOENIX-01 Trial
Acronym: PHOENIX-01
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Administrative barriers
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Juergen Debus, Prof. Dr. Dr. Jürgen Debus, University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHOENIX-01
Record Dates: First submitted 2013-02-18; First posted 2013-02-20 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Locally Advanced Pancreatic Cancer
MeSH Terms: interventions — Heavy Ion Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carbon Ion Radiotherapy (Experimental): Step 1 14 x 3 Gy E 42 Gy E Step 2: 15 x 3 Gy E 45 Gy E Step 3: 16 x 3 Gy E 49 Gy E Step 4: 17 x 3 Gy E 51 Gy E Step 5: 18 x 3 Gy E 54 Gy E
  Interventions: Radiation: Carbon Ion Radiotherapy

INTERVENTIONS:
Radiation: Carbon Ion Radiotherapy — Step 1 14 x 3 Gy E 42 Gy E Step 2: 15 x 3 Gy E 45 Gy E Step 3: 16 x 3 Gy E 49 Gy E Step 4: 17 x 3 Gy E 51 Gy E Step 5: 18 x 3 Gy E 54 Gy E

SUMMARY:
The physical and biological properties of the carbon ion beam promise to improve the therapeutic ratio in patients with pancreatic cancer: Due to the inverted dose profile dose deposition in the entry channel of the beam leads to sparing of normal tissue; the Bragg peak can be directed into the defined target volume, and the sharp dose fall-off thereafter again spares normal tissue behind the target volume. The higher RBE of carbon ions, which has been shown also for pancreatic cancer cell lines in the preclinical setting, is likely to contribute to an increase in local control, and perhaps in OS. Early data from Japanese centers have shown convincing results. The PHOENIX-01 trial is the first trial to evaluate actively delivered carbon ion beams in patients with locally advanced pancreatic cancer within a dose-escalation strategy.

ELIGIBILITY:
Inclusion criteria

Patients meeting all of the following criteria will be considered for admission to the trial:

* histologically confirmed locally advanced pancreatic cancer or imaging defined pancreatic cancer combined with elevated CA-19-9
* macroscopic tumor after biopsy
* age ≥ 18 years of age
* Karnofsky Performance Score >=60
* For women with childbearing potential, (and men) adequate contraception (sexual abstinence, estrogen- or gestagen containing contraceptive medication etc.)
* Female participants: No pregnancy present (pregnancy test required)
* Ability of subject to understand character and individual consequences of the clinical trial
* Written informed consent (must be available before enrolment in the trial)

Exclusion criteria:

Patients presenting with any of the following criteria will not be included in the trial:

* distant metastases
* refusal of the patients to take part in the study
* previous radiotherapy of the abdomen
* Patients who have not yet recovered from acute toxicities of prior therapies
* Known carcinoma < 5 years ago (excluding Carcinoma in situ of the cervix, basal cell carcinoma, squamous cell carcinoma of the skin) requiring immediate treatment interfering with study therapy
* Pregnant or lactating women
* Participation in another clinical study or observation period of competing trials, respectively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2018-05-01 (Estimated)

PRIMARY OUTCOMES:
Acute toxicity of carbon ion radiotherapy observed within 3 months of study treatment | 3 months
  Acute toxicity of carbon ion radiotherapy observed within 3 months of study treatment

SECONDARY OUTCOMES:
imaging response | 2 years
progression-free survival | 2 years
  progression-free survival
overall survival | 2 years
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Heidelberg, Radiation Oncology, Heidelberg, Germany

REFERENCES:
- [Derived] Combs SE, Habermehl D, Kieser M, Dreher C, Werner J, Haselmann R, Jakel O, Jager D, Buchler MW, Debus J. Phase I study evaluating the treatment of patients with locally advanced pancreatic cancer with carbon ion radiotherapy: the PHOENIX-01 trial. BMC Cancer. 2013 Sep 14;13:419. doi: 10.1186/1471-2407-13-419. PMID 24034562